CLINICAL TRIAL: NCT05573945
Title: Developmental Family Centred Care Program in Neonatal Intensive Care Unit
Brief Title: Developmental Care Program in Neonatal Intensive Care Unit
Acronym: CIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Pisa (Other)
Collaborators: Azienda Ospedaliero, Universitaria Pisana (Other); IRCCS Fondazione Stella Maris (Other)
Responsible Party: Principal Investigator, Andrea Guzzetta, Full Professor, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CIN
Record Dates: First submitted 2022-09-15; First posted 2022-10-10 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-01

CONDITIONS: Premature Birth
Keywords: Family-Centered Care; Neonatology; Early intervention; Counseling
MeSH Terms: conditions — Premature Birth | interventions — Sex Education

STUDY DESIGN:
Intervention Model Description: Two intervention groups, Randomised Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Double (Investigator, Outcomes Assessor) Investigator and Outcomes assessors are blind to the group assignment of the infant. Care provider (Parents and Research staff supporting parents in intervention can not be masked to the group assignment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Family Education Only (Experimental): Family Education Only. Parents will be asked to participate in an evidence based program s that includes 6-8 visits with a a trained healthcare provider.
  This program of early intervention based on the promotion of the parent-child relationship through the recognition of behavioral states, methods of interaction, facilitation strategies in the relationship.
  Active listening Visits includes a cycle of 5-6 consecutive meetings lasting about an hour. The meetings will take place in a defined and dedicated space (private room) or if possible (if no other parents are present) at the baby's cradle. The meeting will take place between a single parent and a trained direct operator. This is not a psychotherapeutic intervention but a support that is provided to the parent. The support is mainly based on active listening, on the problems posed by the parent and on the subject's empowerment.
  Interventions: Behavioral: Family Education and Active Listening
- Family Education and Active Listening (Active Comparator): Family Education and Active Listening. Parents of infants will be asked to participate in an evidence based program for parents of NICU infants that includes 6-8 visits with a a trained healthcare provider operator.
  This evidence-based program of early intervention based on the promotion of the parent-child relationship through the recognition of behavioral states, methods of interaction, facilitation strategies in the relationship.
  The program takes its conceptual basis from the Mother Infant Transaction Program (MITP).
  It involves about 6 meetings (1-2 a week) of 30-45 minutes that are carried out during the hospitalisation in the NICU directly at the child's bed between the operator and one or both parents.
  Interventions: Behavioral: Family Education

INTERVENTIONS:
Behavioral: Family Education and Active Listening — Bedside intervention directly with infant with trained healthcare providers and parents. Includes family education meetings completed with individual infant parent/s and trained operator. In addition, weekly meetings of parent/s with a psychologist in a private location for an active listening counselling session.
  Other Names: Intervention A
  Arms: Family Education Only
Behavioral: Family Education — Bedside intervention directly with infant with trained healthcare providers and parents. Includes family education meetings completed with individual infant parent/s and trained operator.
  Other Names: Intervention B
  Arms: Family Education and Active Listening

SUMMARY:
This project is a Randomised Clinical Trial that includes a family centred education intervention and/or non-directive active listening counselling intervention with families of preterm infants at risk for sensori-motor disorders.

DETAILED DESCRIPTION:
Preterm babies, specifically with gestational age < 33+6 weeks, will be recruited and assigned (randomized) into an a Family Education + Active Listening Group (intervention A) or a Family Education Only Group (intervention B).

When the clinical condition of the child is stable the parents are approached for consent and randomised.

All families (in intervention A and intervention B) will receive the evidence-based program of Family Education which is based on the promotion of the parent-child relationship through the recognition of behavioral states, methods of interaction, facilitation strategies in the relationship.

It takes its conceptual basis from the Mother Infant Transaction Program (MITP). It is a specific and re-adapted version for the preterm infant hospitalized in NICU The family education sessions involve about 6 meetings (1-2 a week) of 30-45 minutes that are carried out during the hospitalization in the NICU directly at the child's bed between the operator and one or both parents. Each meeting involves the discussion of one of the following topics.

The Families in intervention group A will also receive 4-6 weekly meetings with a psychologist for an active listening counselling session.

ELIGIBILITY:
Inclusion Criteria:

* Parents of preterm <34 weeks without brain lesion

Exclusion Criteria:

* Parents of infants with brain Lesions
* Parents of clinically unstable infants, based on standard medical evaluation of preterm infants (eg: children with mechanical ventilation or under sedation)
* Parents of infants with genetic-malformative conditions
* Parents with severe psychiatric disorders

Ages: 1 Week to 10 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Parent Infant interaction behaviours coding | 1 months corrected age
  Video footage of key vocal, facial, and motor parental and infant interactive behaviours are analysed using micro coding system.
Parent Infant interaction behaviours coding | 3 months corrected age
  Video footage of key vocal, facial, and motor parental and infant interactive behaviours are analysed using micro coding system.
Parent Infant interaction behaviours coding | 6 months corrected age
  Video footage of key vocal, facial, and motor parental and infant interactive behaviours are analysed using micro coding system.
Developmental outcome assessment | 12 months corrected age
  Bayley Scales of Infant Development Third Edition will be conducted including the Cognitive, Language (Receptive & Expressive), Motor (Gross & Fine), Social-Emotional and Adaptive sub scales. Each sub scale score will be calculated based on the age (months of age) of the infant at the time assessment. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Family well-being questionnaires | Before discharge from the Neonatal Unit (on average at 5 weeks post term age), 3, 6, 12 months corrected age
  The Infant Toddler Quality of Life QuestionnaireTM (ITQOL)
Family well-being questionnaire | Before discharge from the Neonatal Unit (on average at 5 weeks post term age), 3, 6, 12 months corrected age
  Edinburg Postnatal Depression Scale (EPDS)
Family well-being questionnaire | Frame: Before discharge from the Neonatal Unit (on average at 5 weeks post term age), 3, 6, 12 months corrected age
  Depression Anxiety Stress Scale (DASS-21)
Family well-being questionnaire | Before discharge from the Neonatal Unit (on average at 5 weeks post term age), 3, 6, 12 months corrected age
  Coping Orientation to Problems Experienced (COPE - NVI)

OTHER OUTCOMES:
General Movements (GM) | 10-16 weeks corrected age
  The General Movements Assessment (GMA), an observation of infant spontaneous movements will be completed and scored based on a standard protocol of GMA. The observation allows for the understanding of the neurological risk category for neuromotor difficulties.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Stella Maris, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the Individual Participant Data